CLINICAL TRIAL: NCT03826264
Title: a Multinational Multicenter Prospective Transpacific TAVR Registry
Brief Title: Transpacific TAVR Registry
Acronym: TP-TAVR
Status: Recruiting | Type: Observational
Sponsor: Duk-Woo Park, MD (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Duk-Woo Park, MD, Professor, Asan Medical Center, University of Ulsan College of Medicine, Seoul, Korea, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2019-01
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Heart Valve Diseases; Aortic Valve Insufficiency
Keywords: TAVR; TAVI; real-world
MeSH Terms: conditions — Heart Valve Diseases; Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Korea Centers: Seoul, Korea All Patients undergoing TAVR
  Interventions: Procedure: TAVR
- Stanford University: California, USA All Patients undergoing TAVR
  Interventions: Procedure: TAVR
- Northwestern University: Evanston, Illinois, USA All Patients undergoing TAVR
  Interventions: Procedure: TAVR
- Cheng-Hsin Hospital: Taipei, Taiwan All Patients undergoing TAVR
  Interventions: Procedure: TAVR

INTERVENTIONS:
Procedure: TAVR — transcatheter aortic valve replacement (TAVR)

SUMMARY:
This registry evaluates the long-term outcome of Transcatheter aortic valve replacement (TAVR) in real-world clinical practice.

DETAILED DESCRIPTION:
This study is connected with Asian TAVR registry(NCT02308150). Some subjects from Asian TAVR registry continue 10 years follow-up on this TP-TAVR registry.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing TAVR
* Informed consent

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing TAVR
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
Event rate of all cause death | 1 year

SECONDARY OUTCOMES:
Event rate of cardiovascular death | 10 years
  A. Death due to proximate cardiac cause B. Death caused by non-coronary vascular condition C. All procedure-related death D. All valve-related death E. Sudden or unwitnessed death F. Death of unknown cause
Event rate of myocardial infarction | 10 years
  according to Valve Academic Research Consortium (VARC) criteria
Event rate of cerebrovascular accident | 10 years
  stroke and TIA (Transient Ischemic Attack)
Event rate of bleeding | 10 years
  according to Valve Academic Research Consortium (VARC) criteria
Event rate of Vascular access site and access-related complication | 30 days
  according to Valve Academic Research Consortium (VARC) criteria
Event rate of Acute kidney injury | 30 days
Event rate of Permanent pacemaker insertion | 10 years
Event rate of Other TAVR-related complication | 10 years
  A. Conversion to open surgery B. Coronary obstruction C. Mitral valve apparatus damage or dysfunction D. Cardiac tamponade E. Endocarditis F. Valve thrombosis G. Valve mal-positioning H. TAV-in-TAV deployment
Event rate of Prosthetic valve dysfunction | 10 years
  according to Valve Academic Research Consortium (VARC) criteria
  A. Prosthetic aortic valve stenosis B. Prosthesis-patient mismatch C. Prosthetic aortic valve regurgitation
Event rate of Composite endpoint | 10 years
  A. Device success
  B. Early safety
  : death, cerebrovascular event, fatal bleeding, acute kidney injury, coronary obstruction requiring intervention, major vascular complication, valve dysfunction requiring intervention
  C. Clinical efficacy : death, cerebrovascular event, valve-related symptom requiring hospitalization or devastating heart failure, NYHA class* III, IV dyspnea, valve dysfunction
  *the New York Heart Association (NYHA) Functional Classification
Event rate of Structural valve deterioration | 10 years
NYHA class | 30 days
NYHA class | 1 year
Valve area | 1 year
Event rate of free from atrial fibrillation | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan Ching Yuen Yeung, MD, Principal Investigator — Stanford University; James D. Flaherty, MD, Principal Investigator — Northwestern University
Locations (7):
- United States (2):
  - Stanford University, Stanford, California
  - Northwestern Memorial Hospital, Chicago, Illinois
- Second Affiliated Hospital of Zhejiang University, Hangzhou, China
- South Korea (4):
  - Bucheon Sejong Hospital, Bucheon-si
  - Chungnam National University Hospital, Daejeon
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim M, Kang DY, Ahn JM, Kim JB, Yeung AC, Nishi T, Fearon WF, Cantey EP, Flaherty JD, Davidson CJ, Malaisrie SC, Kim HJ, Lee J, Park J, Kim H, Cho S, Choi Y, Park SJ, Park DW. Sex-Specific Disparities in Clinical Outcomes After Transcatheter Aortic Valve Replacement Among Different Racial Populations. JACC Asia. 2024 Feb 13;4(4):292-302. doi: 10.1016/j.jacasi.2023.11.016. eCollection 2024 Apr. PMID 38660112
- [Derived] Kim H, Kang DY, Ahn JM, Kim JB, Yeung AC, Nishi T, Fearon WF, Cantey EP, Flaherty JD, Davidson CJ, Malaisrie SC, Kim N, Kim M, Lee J, Park J, Choi Y, Park SJ, Park DW. Race-Specific Impact of Conventional Surgical Risk Score on 1-Year Mortality After Transcatheter Aortic Valve Replacement. JACC Asia. 2023 Feb 28;3(3):376-387. doi: 10.1016/j.jacasi.2022.11.007. eCollection 2023 Jun. PMID 37323869
- [Derived] Kang DY, Ahn JM, Kim JB, Yeung A, Nishi T, Fearon W, Cantey EP, Flaherty JD, Davidson CJ, Malaisrie SC, Park SY, Yun SC, Ko E, Park H, Lee SA, Kim DH, Kim HJ, Kim JB, Choo SJ, Park DW, Park SJ. Inter-racial differences in patients undergoing transcatheter aortic valve implantation. Heart. 2022 Sep 12;108(19):1562-1570. doi: 10.1136/heartjnl-2021-320364. PMID 35110384
- [Derived] Park H, Ahn JM, Kang DY, Kim JB, Yeung AC, Nishi T, Fearon WF, Cantey EP, Flaherty JD, Davidson CJ, Malaisrie SC, Kim S, Yun SC, Ko E, Lee SA, Kim DH, Kim HJ, Kim JB, Choo SJ, Park DW, Park SJ. Racial Differences in the Incidence and Impact of Prosthesis-Patient Mismatch After Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2021 Dec 27;14(24):2670-2681. doi: 10.1016/j.jcin.2021.08.038. Epub 2021 Nov 24. PMID 34838464